CLINICAL TRIAL: NCT02866097
Title: Strengthening the Delivery of Integrated Community Case Management (iCCM) in Two Districts of Eastern Province, Zambia
Brief Title: Integrated Community Case Management Study in Eastern Province, Zambia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zambia Center for Applied Health Research and Development (Other)
Collaborators: UNICEF (Other); Bill and Melinda Gates Foundation (Other); Boston University (Other); Ministry of Health, Zambia (Other Government); Ministry of Community Development, Mother and Child Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4980/A0/04/001/010
Record Dates: First submitted 2015-12-10; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Malaria; Diarrhea; Pneumonia
Keywords: integrated community case management; Mobile Health (mHealth); rapid diagnostic test; artemether-lumefantrine; amoxicillin; zinc; oral rehydration solution (ORS); District Health Information System 2 (DHIS2); iCCM-DHIS2; ZCAHRD
MeSH Terms: conditions — Malaria; Diarrhea; Pneumonia; Osteoarthritis | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): mHealth inventory management and referrals via text messaging plus supportive supervision of CHWs via an mHealth strategy
  Interventions: Other: mHealth inventory management; Other: Supportive supervision
- Control (Placebo Comparator): ICCM current standard of care with CHWs operating under standard conditions without enhanced inventory management or supportive supervision by mHealth
  Interventions: Other: ICCM current standard of care

INTERVENTIONS:
Other: mHealth inventory management — Improved stock management of iCCM commodities using the DHIS2 mHealth platform
  Other Names: intervention
  Arms: Intervention
Other: Supportive supervision — Strengthening of supportive supervision using DHIS2
  Other Names: intervention
  Arms: Intervention
Other: ICCM current standard of care — ICCM implementation as per current practice without mHealth interventions
  Other Names: Control
  Arms: Control

SUMMARY:
This study will provide important evidence to the Ministry of Community Development, Mother and Child Health (MCDMCH) and the Ministry of Health (MOH) on how to effectively implement iCCM with a focus on improving both the flow of supplies to CHWs as well as the quality of their supervision and mentorship. The overall aim will be to determine whether improvements in supplies for community health workers (CHWs) and strengthened supervision result in improved early and appropriate treatment for children with malaria, pneumonia, and diarrhea in rural Zambia when compared to CHWs offering iCCM without this logistics and supervision support.

DETAILED DESCRIPTION:
The main objective of this study is to strengthen the delivery of integrated community case management (iCCM) of malaria, diarrhea, and pneumonia in Chadiza and Chipata Districts of Eastern Province, through mHealth supported improved supply chain management of iCCM commodities and enhanced supportive supervision of iCCM-trained CHWs.

ELIGIBILITY:
Inclusion Criteria:

* Age <5 years
* Treatment for an iCCM condition (malaria, pneumonia, or diarrhea) by a CHW
* Willingness of the child's caregiver to provide informed consent

Exclusion Criteria:

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3840 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Composite percentage of children appropriately treated for malaria, diarrhea, and pneumonia. | Through study completion, up to six months
  Defined as percentage of sick children under five years of age presenting with an i-CCM condition to an i-CCM trained health worker (CHW or a CHA) who received appropriate treatment for an iCCM condition (composite indicator):
  Appropriate treatment for malaria: received artemisinin-based combination therapy (ACT) for malaria for at least three days or Appropriate treatment for pneumonia: received amoxicillin for pneumonia for at least five days or Appropriate treatment for diarrhea: received zinc in addition to fluid from ORS packet or oral rehydration solution (ORS) liquid or homemade fluid for diarrhea

SECONDARY OUTCOMES:
a) Medicine availability (artemether-lumefantrine) | Through study completion, up to six months
  Defined as percentage of iCCM sites with artemether-lumefantrine in stock during the monthly assessments
b) Clinical supervision coverage | Through study completion, up to six months
  Defined as proportion of CHWs who received at least one supervisory contact (in person) every 3 months during which a sick child visit or scenario was assessed and coaching provided.
c) Virtual supervision coverage (via mobile technology) | Through study completion, up to six months
  Defined as proportion of CHWs who received at least SMS per month from their supervisor reinforcing the appropriate use of the iCCM algorithm for classification and treatment.
d) Average cost per iCCM contact | Through study completion, up to six months
  Defined as average expenditure per iCCM contact by type of condition
e) Diagnostic availability | Through study completion, up to six months
  Defined as percentage of iCCM sites with all iCCM diagnostics (malaria rapid diagnostic tests) in stock during the monthly assessments
f) Medicine availability (amoxicillin) | Through study completion, up to six months
  Defined as percentage of iCCM sites with amoxicillin in stock during the monthly assessments
g) Medicine availability (ORS) | Through study completion, up to six months
  Defined as percentage of iCCM sites with ORS in stock during the monthly assessments
h) Medicine availability (Zinc) | Through study completion, up to six months
  Defined as percentage of iCCM sites with Zinc in stock during the monthly assessments

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Biemba, MBChB, M.Sc, Principal Investigator — ZCAHRD and Boston University; David Hamer, MD, Principal Investigator — Boston University; Boniface M Chiluba, B.Sc, M.Sc, Study Director — Zambia Center for Applied Health Research and Development
Locations (1):
- Chadiza and Chipata Districts, Chipata, Eastern Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the data available to outside parties upon receipt of an appropriate request detailing specific aims and an acceptable analysis plan.

REFERENCES:
- [Derived] Biemba G, Chiluba B, Yeboah-Antwi K, Silavwe V, Lunze K, Mwale RK, Hamer DH, MacLeod WB. Impact of mobile health-enhanced supportive supervision and supply chain management on appropriate integrated community case management of malaria, diarrhoea, and pneumonia in children 2-59 months: A cluster randomised trial in Eastern Province, Zambia. J Glob Health. 2020 Jun;10(1):010425. doi: 10.7189/jogh.10.010425. PMID 32509293